CLINICAL TRIAL: NCT00350987
Title: Procalcitonin Guided Antibiotic Therapy and Hospitalisation in Patients With Lower Respiratory Tract Infections: The "ProHOSP" Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EKBB87/06
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Lower Respiratory Tract Infection; Pneumonia; Bronchitis
Keywords: Procalcitonin, guidelines, LRTI, non-inferiority; COLD
MeSH Terms: conditions — Pneumonia; Bronchitis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- PCT (Experimental): PCT guidance
  Interventions: Behavioral: a strategy based on PCT guided AB therapy
- Guidelines (Active Comparator): enforced guidelines
  Interventions: Behavioral: a strategy based on PCT guided AB therapy

INTERVENTIONS:
Behavioral: a strategy based on PCT guided AB therapy — In this study a strategy based on PCT guided AB therapy with enforced guideline implementation will be compared.

SUMMARY:
The aim of this study is to test if procalcitonin (PCT) guided antibiotic stewardship in patients with lower respiratory tract infection (LRTI) will be non-inferior, with at worst a 7.5% higher combined failure rate, as compared to standard care practice (current guidelines for LRTI) with reduced total antibiotic (AB) use and hospitalization rate and duration, respectively.

DETAILED DESCRIPTION:
Background: Acute lower respiratory tract infections (LRTI), i.e. acute bronchitis and acute exacerbations of chronic obstructive pulmonary disease (AECOPD), and community-acquired pneumonia (CAP), employ important hospital resources and often unnecessary antibiotic (AB) treatment courses. We demonstrated in four intervention trials enrolling > 1200 patients that procalcitonin (PCT)-guidance markedly reduces AB prescription and duration. To ascertain the external validity, safety and potential to improve the allocation of health care resources, a non-inferiority multicenter intervention trial has to be done.

Aim: To compare a strategy based on evidence-based guidelines with PCT guided AB therapy in LRTI with respect to outcome (combined disease-specific failure rates), use of AB and hospital resources.

Design: Investigator-initiated, controlled trial with an open intervention. Patients admitted with LRTI to hospital will be included and randomized 1:1 either to standard management or to the PCT-guided prescription of AB. Randomization will be stratified by centre (the hospital) and type of LRTI (Acute bronchitis/AECOPD/CAP).

Setting: Teaching hospitals and tertiary care clinics from northwestern and central Switzerland.

Patients: 18 years or older, with LRTI of > 1 and < 28 days duration. Excluded are patients without informed consent, not fluent in German, unlikely to comply, severe immuno-suppression, terminal condition where death is expected to occur during the current hospitalization, immediate need for intensive care.

Endpoints:

* Primary: Risk of combined disease-specific failure after 30 days.
* Secondary: AB exposure, side effects from ABs, time to AB treatment, rate and duration of hospitalization, time to clinical stability, disease activity scores.

Endpoints will be assessed at baseline, daily in hospitalized patients and after 30 and 180 days by structured phone interviews by blinded medical students.

Intervention: Participating physicians will receive evidence-based guidelines for the management of patients with LRTIs. Patients with LRTI will be randomized to PCT plus guidelines ("PCT group") versus only guidelines-guided AB treatment ("control group"). In patients randomized to the PCT group the use of ABs will be more or less discouraged (< 0.1 or < 0.25 ug/L) or encouraged (> 0.5 or > 0.25 ug/L), respectively. A re-evaluation after 6 to 24 hours in patients in whom antibiotics are withheld with worsening or non-improvement of vital signs with PCT (< 0.1 or < 0.25 ug/L) is recommended. During hospitalization, patients with AB treatment will be reassessed at day 3, 5 and 7 and in patients randomized to the PCT group it is recommended to stop AB based on PCT levels. In AB-treated outpatients or discharged patients with AECOPD and CAP randomized to the PCT group with uncomplicated course, the recommended duration of AB therapy will be based on the last PCT level and will be as follows: > 0.5 ug/L, 5 days; > 0.25 ug/L, 3 days; < 0.25 ug/L, stop AB.

Variables and measurement: Centers have to consecutively enroll all patients with LRTI. Baseline data on medical history and clinical items, additional diagnostic tests, co-morbidity, final prescribed treatment and reasons for hospital admission and stay will be collected. After a pilot/feasibility phase of 3 months, study recruitment will continue from Mar 2007 to Apr 2008.

Study hypothesis: PCT guidance will be non-inferior with at worst a 7.5% higher combined failure rate as compared to standard care practice with a reduced total AB use and hospitalization rate and duration, respectively.

Analyses: These will be done based on an intention-to-treat and a per-protocol principle. With an assumed combined failure rate of 15% to 20%, a non-inferiority margin of 7.5%, a maximum of 5% losses to follow-up, a value of 5% and power of 90%, the total sample size is 806 α one-sided to 1002.

Interim monitoring: Regular review of serious adverse events, quality and integrity of the study by an independent data safety and monitoring board. Safety interim analysis and blinded assessment (i.e., with both arms pooled) of the diagnostic and prognostic accuracy of biomarkers after 50% of the patients recruited.

Ancillary projects: Six related projects will be performed alongside to this study (including, cost-effectiveness, nursing and social influence on hospitalization, prognostic value of novel biomarkers) to synergize scientific efforts.

Significance: Due to the high prevalence and absorption of hospital resources, this study will offer the potential for large improvements in the management of LRTIs, along with substantial reduction in hospitalization costs and AB resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older, admitted from the community or a nursing home with acute (i.e., at least 1 day but less than 28 days) LRTI as the main diagnosis consisting of having at least two of the following:

   * new or increased respiratory signs or symptoms (i.e., cough, sputum production, dyspnea, auscultatory findings of abnormal breath sounds and rales, pleuritic chest pain) with or without inflammatory signs (core body temperature > 38.0° C, leukocyte count > 10 or < 4 x 10^9 cells L-1).
   * CAP is defined by the presence of LRTI along with a new or increased infiltrate on chest radiograph. Severity scores of CAP (pneumonia severity index [PSI] and CURB-65) will be calculated.
   * COPD is defined by post-bronchodilator spirometric criteria according to the GOLD-guidelines as a FEV1/FVC ratio below 70% and the severity categorized into mild (FEV1 <= 80% of predicted), moderate (50% >= FEV1 < 80%), severe (30% >= FEV1 < 50%) and very severe (FEV1 < 30%), respectively. Severity of acute exacerbations of COPD will be graded as proposed. Acute bronchitis is defined as LRTI in the absence of an underlying lung disease or focal chest signs and infiltrates on chest X-ray, respectively. Patients who are on admission judged as having an LRTI but have another final diagnosis, will be classified as "others".
2. Ability to understand verbal and written instructions and informed consent.

Exclusion Criteria:

1. Patients unable to give written informed consent, e.g. with severe dementia or patients not understanding German (or other local language) and no translation (e.g. family members) available.
2. Patients with active intravenous drug use.
3. Severe immunosuppression (e.g. patients infected with human immunodeficiency virus infection and a CD4 count below 350 x 10^9/L, patients on immunosuppressive therapy after solid organ transplantation and neutropenic patients with present neutrophil count < 500 x 10^9/L and patients under chemotherapy with neutrophils 500-1000 x 10^9/L with an expected decrease to values < 500 x 10^9/L); patients with cystic fibrosis, infection with M. tuberculosis, L. pneumophila, Listeria spp. hospital stay within 14 days of inclusion.
4. Accompanying chronic (e.g. osteomyelitis), abscess (e.g. brain, pleural empyema) infection or endocarditis.
5. Terminal and very severe medical co-morbidity where death is imminent or has to be expected in the current hospitalization (e.g. due to malignancy, cardiac, renal or hepatic failure, comfort therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
the risk of disease specific failure | within 1 month COPD

SECONDARY OUTCOMES:
time to AB treatment/prescription rate, duration, rate and doses, first change, side-effects, hospitalization and discharge
clinical stability, disease activity score, restriction days, function/health state, prediction rules and diagnostic and prognostic accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Mjriam Christ-Crain, Dr.med., Principal Investigator — University Hospital in Basel; Philipp Schuetz, Dr.med., Principal Investigator — University Hospital in Basel; Werner Zimmerli, Prof., Principal Investigator — University Hospital in Liestal, Switzerland; Beat Mueller, Prof., Study Director — University Hospital in Basel
Locations (1):
- University Hospital in Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Result] Christ-Crain M, Morgenthaler NG, Stolz D, Muller C, Bingisser R, Harbarth S, Tamm M, Struck J, Bergmann A, Muller B. Pro-adrenomedullin to predict severity and outcome in community-acquired pneumonia [ISRCTN04176397]. Crit Care. 2006;10(3):R96. doi: 10.1186/cc4955. Epub 2006 Jun 28. PMID 16805922
- [Result] Christ-Crain M, Stolz D, Bingisser R, Muller C, Miedinger D, Huber PR, Zimmerli W, Harbarth S, Tamm M, Muller B. Procalcitonin guidance of antibiotic therapy in community-acquired pneumonia: a randomized trial. Am J Respir Crit Care Med. 2006 Jul 1;174(1):84-93. doi: 10.1164/rccm.200512-1922OC. Epub 2006 Apr 7. PMID 16603606
- [Result] Briel M, Christ-Crain M, Young J, Schuetz P, Huber P, Periat P, Bucher HC, Muller B. Procalcitonin-guided antibiotic use versus a standard approach for acute respiratory tract infections in primary care: study protocol for a randomised controlled trial and baseline characteristics of participating general practitioners [ISRCTN73182671]. BMC Fam Pract. 2005 Aug 18;6:34. doi: 10.1186/1471-2296-6-34. PMID 16107222
- [Result] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884
- [Derived] Schuetz P, Wolbers M, Christ-Crain M, Thomann R, Falconnier C, Widmer I, Neidert S, Fricker T, Blum C, Schild U, Morgenthaler NG, Schoenenberger R, Henzen C, Bregenzer T, Hoess C, Krause M, Bucher HC, Zimmerli W, Mueller B; ProHOSP Study Group. Prohormones for prediction of adverse medical outcome in community-acquired pneumonia and lower respiratory tract infections. Crit Care. 2010;14(3):R106. doi: 10.1186/cc9055. Epub 2010 Jun 8. PMID 20529344
- [Derived] Muller F, Christ-Crain M, Bregenzer T, Krause M, Zimmerli W, Mueller B, Schuetz P; ProHOSP Study Group. Procalcitonin levels predict bacteremia in patients with community-acquired pneumonia: a prospective cohort trial. Chest. 2010 Jul;138(1):121-9. doi: 10.1378/chest.09-2920. Epub 2010 Mar 18. PMID 20299634
- [Derived] Baehni C, Meier S, Spreiter P, Schild U, Regez K, Bossart R, Thomann R, Falconnier C, Christ-Crain M, De Geest S, Muller B, Schuetz P; ProHOSP Study Group. Which patients with lower respiratory tract infections need inpatient treatment? Perceptions of physicians, nurses, patients and relatives. BMC Pulm Med. 2010 Mar 11;10:12. doi: 10.1186/1471-2466-10-12. PMID 20222964